CLINICAL TRIAL: NCT07283991
Title: Prospective Single-Arm Study of QL1706 Plus Chemotherapy for Borderline Resectable Esophageal Cancer
Brief Title: QL1706 Plus Chemotherapy for Borderline Resectable Esophageal Cancer
Acronym: BRICES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of Department of Thoracic Surgery, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-028; MR-31-25-068250 (Registry Identifier: MR-31-25-068250)
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aparolitolovureli plus chemotherapy group (Experimental)
  Interventions: Drug: chemotherapy combined with Aparolitolovureli immunotherapy

INTERVENTIONS:
Drug: chemotherapy combined with Aparolitolovureli immunotherapy — After enrollment, patients will receive first-stage treatment consisting of cisplatin plus nanoparticle albumin-bound paclitaxel chemotherapy combined with Aparolitolovureli immunotherapy for 2 to 4 cycles. If the tumor is assessed as resectable, radical esophagectomy will be performed. If the tumor remains unresectable, definitive concurrent chemoradiotherapy will be administered. Following radical esophagectomy, patients will enter the second stage of treatment with Aparolitolovureli maintenance immunotherapy for up to 1 year (a maximum of 14 cycles during the maintenance phase).

SUMMARY:
China bears a disproportionately high burden of esophageal cancer, accounting for approximately 50% of newly diagnosed cases worldwide, with an average 5-year survival rate of only 30%. Esophageal adenocarcinoma and squamous cell carcinoma (ESCC) are the major pathological subtypes, among which squamous cell carcinoma predominates in Asian populations. More than 90% of esophageal cancer cases in China are ESCC.

Optimal treatment for locally advanced esophageal cancer remains a matter of debate. Findings from Japanese clinical studies such as JCOG1109 have demonstrated that neoadjuvant chemotherapy can significantly improve long-term survival in patients with locally advanced ESCC. Neoadjuvant chemotherapy followed by surgery has therefore become one of the preferred treatment strategies.

Preclinical evidence suggests synergistic interactions between chemotherapy and immunotherapy, potentially enhancing treatment efficacy. Moreover, clinical trials such as ESCORT-NEO and NCCES01 have validated the safety and effectiveness of immunochemotherapy for locally advanced esophageal cancer. Consequently, chemotherapy combined with immunotherapy has emerged as a promising approach for improving survival outcomes in this patient population.

A Phase II clinical trial involving the investigational drug Aparolitolovureli was conducted in 39 patients with unresectable locally advanced ESCC, evaluating a regimen of radical chemoradiotherapy combined with immunotherapy followed by Aparolitolovureli maintenance. The study reported a median progression-free survival (mPFS) of 13.99 months, with 12-month PFS and OS rates of 62.1% and 86.2%, respectively, demonstrating encouraging efficacy. These results, together with supporting preclinical data, suggest that immunochemotherapy is both feasible and effective in locally advanced esophageal cancer.

Based on this foundation, our research team proposes a single-arm clinical study in patients with borderline resectable locally advanced ESCC. A total of 24 participants will receive 2-4 cycles of inductive immunochemotherapy with Aparolitolovureli plus cisplatin and paclitaxel. Patients deemed resectable after reassessment will undergo radical esophagectomy, followed by Aparolitolovureli maintenance therapy. The study aims to evaluate the efficacy and safety of this treatment strategy and provide scientific evidence and clinical guidance to improve the overall prognosis of patients with ESCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma.
* Clinical stage cT4a, or at least one lymph node suspected of invading adjacent structures, or conglomerated/enlarged lymph nodes, or supraclavicular lymph node metastasis.
* No prior anti-tumor treatment before enrollment.
* Age ≥ 18 years.
* ECOG Performance Status score of 0-1.
* Signed written informed consent.

Exclusion Criteria:

* Presence of autoimmune disease.
* Requiring systemic corticosteroid therapy or other immunosuppressive medications.
* Symptomatic interstitial lung disease.
* Known hypersensitivity to the investigational drug(s).
* Pregnant or breastfeeding women.
* Patients of childbearing potential who refuse to use effective contraception.
* Prior treatment with immune checkpoint inhibitors or any agents targeting T-cell co-stimulatory/co-inhibitory pathways.
* Any condition deemed by the investigator to increase treatment risk or confound study outcome assessment.
* Prior esophageal cancer-related chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | at 2 weeks post-surgery
  R0 resection rate confirmed by pathological evaluation.

SECONDARY OUTCOMES:
major pathological response rate | at 2 weeks post-surgery
  short-term efficacy of the treatment regimen (major pathological response rate) .The proportion of patients achieving major pathological response, as assessed by tumor regression grading on postoperative pathological specimens.
radiological response rate | at 1 months post-treatment
  short-term efficacy of the treatment regimen（radiological) . The objective response rate (complete response + partial response) assessed according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
3-year progression-free survival rate | at 3 years post-treatment
  long-term oncological outcomes (3-year progression-free survival) The proportion of patients alive and free from disease progression within 3 years from the initiation of treatment.
3-year overall survival rate | at 3 years post-treatment
  long-term oncological outcomes (3-year overall survival) . The proportion of patients alive at 3 years from the initiation of treatment, regardless of the cause of death.

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: With publication
Access Criteria: Interested investigators will be required to submit a formal letter of intent outlining research aims, rationale, and approach. Furthermore, documentation of local IRB approval, including a description of type of review, should be submitted with the data request.